CLINICAL TRIAL: NCT01808352
Title: Pre-Exposure Prophylaxis (PrEP) Initiation and Adherence Among Black Men Who Have Sex With Men (BMSM) in Three U.S. Cities
Brief Title: HPTN 073 Black Men Who Have Sex With Men (MSM) Pre-Exposure Prophylaxis (PrEP)
Status: Completed | Type: Observational
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HPTN 073
Record Dates: First submitted 2013-03-05; First posted 2013-03-11 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HIV
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine specimens to be stored after the end of the study for possible future testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Observational study
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — HPTN 073 is an observational study in MSM in the United States

SUMMARY:
Black men who have sex with men (MSM) Pre-Exposure Prophylaxis (PrEP) Study with Client Centered Care Coordination (C4) Component.

DETAILED DESCRIPTION:
An open label demonstration study with PrEP and Client Centered Care Coordination (C4) to assess the initiation, acceptability, safety, and feasibility of PrEP for Black MSM (BMSM) in three US Cities. A subset of participants will also be recruited to participate in qualitative interviews about facilitators and barriers regarding PrEP. The study will recruit HIV-uninfected BMSM at risk for HIV infection in three US Cities. Enrollment will include those aged 18 and over with an effort to recruit an equal number of BMSM under age 25 and over age 25 with a total of 225 participants (75 per site).

ELIGIBILITY:
Inclusion Criteria:

BMSM who meet all of the following criteria are eligible for inclusion in this study:

* 18 years of age or older
* No prior HIV diagnosis (self-report)
* Male at birth
* High risk for acquiring HIV infection including any one of the following in the previous 6 months:

  * Unprotected sex during receptive or insertive anal intercourse with a male partner
  * Any protected or unprotected:

    i. Receptive or insertive anal intercourse with more than three male sex partners ii. Exchange of money, gifts, shelter or drugs for receptive or insertive anal sex with a male partner iii. Receptive or insertive anal sex while under the influence of drugs or alcohol (i.e., high or drunk within two hours of the sex act) according to self-report"
  * STI diagnosis (i.e., syphilis, gonorrhea and chlamydia) by self-report
* Willing to provide locator information in accordance with the Study Specific Procedures (SSP) Manual
* Urine dipstick negative or trace for protein and glucose
* Hemoglobin > 11 g/dL, absolute neutrophil count > 750 cells/mm3, and platelet count ≥ 100,000/mm3
* Serum creatinine < upper limit of normal (ULN) and calculated creatinine clearance of at least 60 mL/min by the Cockcroft-Gault formula where:

  o eCcr in mL/min = [(140 - age in years) x (actual body weight in kg)] / (72 x serum creatinine in mg/dL) Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 3 times the upper limit of normal (ULN)
* Total bilirubin < 2.5 ULN
* Hepatitis B surface antigen (HBsAg) negative

Exclusion Criteria:

BMSM who meet any of the following criteria will be excluded from this study:

* Any reactive or positive HIV test at Screening, even if subsequent testing indicates that the person is HIV-uninfected
* Transgender
* Active or chronic hepatitis B infection (as evidenced by HBsAg, HbsAb, and HbcAb testing)
* Planning to move out of the area or to travel for more than 3 months during the study follow-up period
* Unwilling to adhere to study procedures
* Current participation in any research study via self-report (however, strictly non-HIV centered observational studies are not exclusionary)
* Previous participation in an HIV vaccine study is exclusionary unless documented evidence of enrollment into a placebo arm
* Use of ARV drugs (PrEP or PEP) in the last 60 days
* Prior history of a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract or drug absorption (provided by self-report, or obtained from medical history or records)
* Receipt of prohibited medications: interleukin therapy, medications with significant nephrotoxic potential (including but not limited to amphotericin B, aminoglycosides, cidofovir, foscarnet and systemic chemotherapy), and medications that may inhibit or compete for elimination via active renal tubular secretion (including but not limited to probenecid) - (provided by self-report, or obtained from medical history or medical records)
* Any condition, that in the opinion of study staff, would make participation in the study unsafe, or interfere with achieving the study objective

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-uninfected BMSM at risk for HIV infection in three U.S. cities. Enrollment will include those aged 18 and over with efforts at each site to attempt to recruit an equal number of BMSM under age 25 and 25 and over.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Initiation of PrEP | 30 months
  Documented in either study CRFs or ACASI
Adherence to PrEP | 30 months
  Adherence will be assessed via self-report (ACASI), PBMCs and plasma concentration

SECONDARY OUTCOMES:
Adverse events | 30 months
  Graded via DAIDS Toxicity Grading System determined by review of reported adverse events (clinical and laboratory)
STIs | 30 months
  Rectal and urine GC/CT, and NAAT for syphilis and chlamydia
Changes in sexual risk-taking behavior | 30 months
  Measured by ACASI assessments
Initiate or decline PrEP | 30 months
  Refusal rates will be measured by ACASI assessments
Incident HIV-seroconversions/characteristics | 30 months
  HIV RNA and genotyping will be performed at the NL on samples confirmed to be HIV infected
Participant perception of care and referral plan | 30 months
  Assessed via interviewer-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — UCLA Vice Street Clinic; Manya Magnus, PhD, MPH, Principal Investigator — George Washington University CRS; Lisa Hightow-Weidman, Principal Investigator — UNC CRS
Locations (3):
- United States (3):
  - UCLA Vine Street Clinic, Los Angeles, California
  - George Washington University CRS, Washington D.C., District of Columbia
  - UNC CRS, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hightow-Weidman LB, Magnus M, Beauchamp G, Hurt CB, Shoptaw S, Emel L, Piwowar-Manning E, Mayer KH, Nelson LE, Wilton L, Watkins P, Whitfield D, Fields SD, Wheeler D. Incidence and Correlates of Sexually Transmitted Infections Among Black Men Who Have Sex With Men Participating in the HIV Prevention Trials Network 073 Preexposure Prophylaxis Study. Clin Infect Dis. 2019 Oct 15;69(9):1597-1604. doi: 10.1093/cid/ciy1141. PMID 30615169